CLINICAL TRIAL: NCT02182011
Title: An Open-label, Randomised, Parallel-group Comparison to Investigate the Procoagulant Effect of Tenecteplase (TNK-tPA), Alteplase (Rt-PA) and Streptokinase (SK) Administered to Patients With AMI
Brief Title: A Study to Investigate the Procoagulant Effect of Tenecteplase (TNK-tPA), Alteplase (Rt-PA) and Streptokinase (SK) Administered to Patients With Acute Myocardial Infarction (AMI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1123.5
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Tenecteplase; Tissue Plasminogen Activator; Streptokinase

ARMS (3):
- Tenecteplase (Experimental): Single i.v. bolus followed by infusion, weight adjusted
  Interventions: Drug: Tenecteplase
- Alteplase (Active Comparator): Single i.v. bolus followed by infusion
  Interventions: Drug: Alteplase
- Streptokinase (Active Comparator): I.V. infusion
  Interventions: Drug: Streptokinase

INTERVENTIONS:
Drug: Tenecteplase
  Arms: Tenecteplase
Drug: Alteplase
  Arms: Alteplase
Drug: Streptokinase
  Arms: Streptokinase

SUMMARY:
Primary objective: to evaluate the procoagulant effect of TNK-tPA compared to rt-PA and streptokinase, administered to patients with AMI, by measuring the concentration of TAT at 2 hours after the start of treatment versus baseline values.

Secondary objective: change from baseline in concentration of TAT at 6 and 24 hours; change from baseline in concentration of D-dimers, F1+2, PAI-1, PAP at 2, 6 and 24 hours. Incidence of adverse events (AE's), in -hospital complications, major or minor bleedings and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Onset of symptoms of AMI within 6 hours from randomisation
* A twelve-lead electrocardiogram (ECG) showing ST-segment elevation ≥ 0.1 millivolt (mV) in two or more limb leads, or ≥ 0.2 mV in two or more contiguous precordial leads indicative of AMI, or new left bundle-branch block
* Age ≥ 18

Exclusion Criteria:

* Hypertension defined as blood pressure > 180/110 mmHg (systolic BP > 180 mmHg and/or diastolic BP > 110 mmHg) on repeated measurements during current admission prior to randomisation
* Use of abciximab (ReoPro®) within the preceding 7 days or eptifibatide (Integrilin®) or tirofiban (aggrastat®) within the past 48 hours
* Use of heparin within the preceding 12 hours
* Current therapeutic oral anticoagulation
* Major surgery, biopsy of a parenchymal organ, or significant trauma within 2 months
* Any minor head trauma and any other trauma occurring after the onset of the current myocardial infarction
* Any known history of stroke or transient ischemic attack or dementia
* Any known structural damage of the central nervous system
* Ruptured aortic aneurism
* Active bleeding
* Prolonged cardiopulmonary resuscitation (> 10 minutes) in the previous two weeks
* Pregnancy or lactation, parturition within the previous 30 days. Women of childbearing potential must have a negative pregnancy test
* Any known active participation in another investigative drug study or device protocol in the past 30 days
* Previous enrolment in this study
* Any other condition that the investigator feels would place the patient at increased risk if the investigational therapy were initiated
* Inability to follow the protocol and comply with follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2000-05; Primary Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in concentration of thrombin anti-thrombin complex (TAT) | Baseline, 2 hours after start of treatment

SECONDARY OUTCOMES:
Changes from baseline in TAT | Baseline, 6 and 24 hours after start of treatment
Changes from baseline in D-dimers | Baseline, 2, 6 and 24 hours after start of treatment
Changes from baseline in prothrombin fragments 1+2 (F1+F2) | Baseline, 2, 6 and 24 hours after start of treatment
Changes from baseline in plasminogen-activator inhibitor-1 (PAI-1) | Baseline, 2, 6 and 24 hours after start of treatment
Changes from baseline in plasmin-antiplasmin complex (PAP) | Baseline, 2, 6 and 24 hours after start of treatment
Occurrence of adverse events (AE's) | Up to 30 days
Occurrence of major bleedings | Up to 30 days
Occurrence of minor bleedings | Up to 30 days
Occurrence of serious adverse events (SAE's) | Up to 30 days
Occurrence of in-hospital complications | Start of treatment until discharge from hospital